CLINICAL TRIAL: NCT01818336
Title: Confirmatory Study to Examine Negative Predictive Value (NPV) and Safety of Skin Testing With PRE-PEN, a Minor Determinant MIxture (MDM) of Penicillin Antigens, and Amoxicillin Reagent Against an Oral Challenge With Amoxicillin
Brief Title: Evaluation of Skin Testing Reagents for Penicillin Allergy
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AllerQuest LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: AQ-2010-001; AllerQuest LLC (Other Grant/Funding Number: AQ-2010-001)
Record Dates: First submitted 2013-03-11; First posted 2013-03-26 (Estimated); Results first posted 2017-01-04 (Estimated); Last update posted 2017-01-04 (Estimated); Status verified 2016-11

CONDITIONS: History of IgE Dependent Reaction to a Penicillin Product
Keywords: penicillin allergy
MeSH Terms: interventions — benzylpenicilloyl G polylysine; Penicillin G; benzylpenicilloic acid; Amoxicillin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- all subjects (Experimental): Intervention: Penicillin skin test kit
  Subjects with negative intradermal tests will be given single oral amoxicillin challenge dose and followed for 72 hours for IgE dependent reactions.
  Interventions: Drug: Penicillin skin test kit

INTERVENTIONS:
Drug: Penicillin skin test kit — Allergy skin testing is done by puncture and intradermal. If all tests negative, subjects receive an oral amoxicillin challenge.
  Other Names: PRE-PEN (benzylpenicilloyl polylysine); MDM (minor determinant mixture of penicillins); benzylpenicillin; benzylpenicilloate; benzylpenilloate; amoxicillin

SUMMARY:
A self- or parent-reported history of penicillin allergy excludes approximately 10% of the US population from receiving penicillin (Kerr 1994, Kagy, Blaiss 1998, Solensky et al. 2000, Neugut et al. 2001). Yet approximately 80% of patients labeled as allergic to the penicillins can safely take these antibiotics without fear of a life-threatening reaction (Gadde et al. 1993, Macy et al. 1997). The outcomes of this erroneous classification of patients include unnecessary denial of an effective and well-tolerated class of antibiotics, which are often the treatment of choice.

The primary aim of skin testing with the Penicillin Skin Test Kit is to identify subjects at very low risk of developing acute IgE-dependent reactions when given a penicillin or cross-reacting drug. The negative predictive value (NPV) of skin testing is assessed by oral challenge with a penicillin.

DETAILED DESCRIPTION:
This is a prospective, open-label investigation of skin testing with the Penicillin Skin Test Kit in subjects at least 18 years of age with a self-reported history of possible IgE-dependent penicillin hypersensitivity.

At screening on Day 1, subjects and their parents/legal guardians (if applicable) will sign the informed consent form/ pediatric assent form. Following consent/assent, demographic information and medical history will be obtained, including prior and current medication use. Subjects will also be asked if they have had a respiratory infection in the past 2 weeks or antibiotics within the past 4 weeks. A physical examination will be performed, along with measurements of vital signs and, in subjects >5 years of age with active asthma, peak expiratory flow rate (PEFR). A urine pregnancy test will be obtained for all female subjects of childbearing potential.

The skin test procedure will first involve puncture testing. Skin test reagents will include the Penicillin Skin Test Kit, histamine (positive control), and sodium chloride (negative control). Subjects who have negative skin puncture test results to any of the drug antigens contained within the Penicillin Skin Test Kit will then undergo intradermal testing in duplicate. Subjects who have a positive reaction to one or more puncture or intradermal tests contained within the Penicillin Skin Test Kit will be discharged from the study. However, subjects with any positive skin test to drug antigens in the Penicillin Skin Test Kit will be asked to return for retesting (puncture and intradermal) in 4 weeks.

Subjects who have negative puncture and intradermal test results will be given the oral amoxicillin challenge, which will be comprised of a single, full oral dose of amoxicillin. The purpose of the oral amoxicillin challenge is to confirm lack of allergy and confirm the NPV (Negative Predictive Value) of skin testing. Subjects will be monitored at the study site for 1 hour following oral amoxicillin challenge and then sent home. The study site will follow-up by telephone with all subjects (or their parents/legal guardians in the case of young children) ≥72 hours after administration of the oral amoxicillin challenge.

Adverse events (AEs) will be recorded from administration of the Penicillin Skin Test throughout the 3-day study period as spontaneously reported by subjects or observed by the site staff.

Two normal subjects (i.e., no history of penicillin allergy) will be skin tested at each site to provide data on skin test specificity.

ELIGIBILITY:
Inclusion Criteria:

1. Subject must have provided written, informed consent prior to performance of any procedures.
2. Subject can be male or female and must be generally healthy and at least 18 years of age.
3. Subject must have a reported history of possible IgE dependent reaction to a penicillin or its semi-synthetic derivatives, including one or more of the following: anaphylaxis, decreased blood pressure and/or diminished consciousness, upper or lower airway obstruction, angioedema, urticaria, and/or generalized pruritic rash.

Exclusion Criteria:

1. Subject who has exhibited a systemic allergic reaction to previous skin-test administration of PRE-PEN, MDM, or individual penicillin metabolites (benzylpenicillin, benzylpenicilloate, or benzylpenilloate).
2. Subject who is pregnant or lactating.
3. Subject who has had a respiratory infection within the past 2 weeks or has taken antibiotics of any kind during the past 2 weeks (except for topical antibiotics for acne).
4. Subject who has taken an oral H1-antihistamine within 72 hours prior to skin testing.
5. Subject who has taken hydroxyzine or doxepin within 7 days prior to skin testing.
6. Subject who has had a penicillin reaction, including semisynthetic penicillins, within the last 6 weeks prior to skin testing.
7. Subject who has received an investigational drug within 30 days prior to skin testing or who plans to participate in a study in which an investigational drug will be administered within the 30 days following skin testing.
8. Subjects who have planned hospitalizations or medical or surgical procedures during the 72 hours following the oral amoxicillin challenge.
9. Subjects who plan to take any new prescription or over-the-counter medications or herbal supplements during the 72 hours following the oral amoxicillin challenge.
10. Subject who has had a previous adverse reaction to penicillin or semisynthetic derivative and subsequently tolerated a penicillin or semisynthetic derivative without an adverse experience.
11. Subject who, in the investigator's opinion, has any other social or medical condition (e.g. fever, rash) that may place the subject at increased risk or may confound the interpretation of the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 481 (Actual)
Dates: Start 2012-12; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: N. Franklin Adkinson, Jr., MD, Study Director — AllerQuest LLC
Locations (13):
- United States (13):
  - Alabama Allergy & Asthma Center, Homewood, Alabama
  - Allergy Associates of Tucson, Tucson, Arizona
  - Allergy & Asthma Clinical Research, Walnut Creek, California
  - Fairfield County Allergy, Asthma & Immunology Assoc., Inc., Norwalk, Connecticut
  - Ct. Asthma & Allergy Center LLC, West Hartford, Connecticut
  - Windom Allergy, Sarasota, Florida
  - Atlanta Allergy and Asthma Clinic, Atlanta, Georgia
  - Mayo Clinic, Rochester, Minnesota
  - Washington University Medical School, St Louis, Missouri
  - Midwest Allergy & Asthma Clinic PC, Omaha, Nebraska
  - Corvallis Clinic, Corvallis, Oregon
  - Allergy & Asthma Care, Germantown, Tennessee
  - Northwest Asthma & Allergy Center, Redmond, Washington

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This was a prospective, open-label investigation of skin testing with the Penicillin Skin Test Kit conducted at 13 asthma and allergy centers in the United States.
Pre-assignment Details: 455 History pos subj enrolled + 2 control subj @ 13 centers. All 481 subj were skin tested(ST) and included in safety population. 64 subj (all history pos) had pos or discordant skin tests and were excluded from ITT population of 391(455 - 64). The subset of 59 ST pos subjects were invited back at 4 weeks for repeat ST; 47 ST pos subj returned
Groups:
- Intent-to-Treat Population: All subjects who had valid skin testing performed (i.e., administered all components of the Penicillin Skin Test Kit and the histamine and control results were valid) and who received the oral amoxicillin challenge.
- Subjects in Retest Population: All subjects who initially tested positive to any of the initial skin tests with penicillin reagents and subsequently returned after 4 weeks for retesting.
Period: Overall Study
Arm/Group | Intent-to-Treat Population | Subjects in Retest Population
Started | 391 | 59
Completed | 391 | 47
Not Completed | 0 | 12
Not completed — Declined retest visit | 0 | 11
Not completed — Lost to Follow-up | 0 | 1

BASELINE CHARACTERISTICS:
Population: Total subjects enrolled in the study
Groups:
- Safety Population: All subjects who had skin testing performed (i.e., administered any component of the Penicillin Skin Test Kit).
Arm/Group | Safety Population
Number analyzed (Participants) | 481
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: Safety population is equal to all enrolled subjects. ITT, Per-protocol, and Re-skin tested subpopulations have been defined elsewhere.
  years
    Safety Population | 49.4 (16.34)
    Intent-to-Treat Population: number analyzed (Participants) | 391
    Intent-to-Treat Population | 50.2 (16.40)
    Per-Protocol Population: number analyzed (Participants) | 373
    Per-Protocol Population | 50.2 (16.49)
    Retest Population: number analyzed (Participants) | 59
    Retest Population | 50.5 (15.32)
Gender [Count of Participants; unit: Participants]
  Female | 138
  Male | 343
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 14
  Not Hispanic or Latino | 467
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2
  Asian | 6
  Native Hawaiian or Other Pacific Islander | 1
  Black or African American | 16
  White | 440
  More than one race | 0
  Unknown or Not Reported | 16
Region of Enrollment [Number; unit: participants]
  United States | 481
Penicillin allergy history [Number; unit: participants]
  No | 26
  Yes | 455
Previous penicillin testing history [Number; unit: participants]
  No | 464
  Yes | 17

OUTCOME MEASURES:

1. Primary Outcome: Negative Predictive Value
Description: The primary endpoint was the negative predictive value (NPV), which was estimated as p = percentage of n history-positive subjects with negative skin tests from the Penicillin Allergy Skin Test Kit (as confirmed with an overall negative result for the skin puncture/intradermal testing) who do not experience an IgE-dependent hypersensitivity reaction within 72 hours of the oral amoxicillin challenge.
Time Frame: 72 hours
Population: The Intent-to-Treat Population; all subjects with valid skin testing performed (ie, administered all components of the penicillin skin test kit and the histamine/control results were valid), who had negative intradermal skin tests with all 3 Kit reagents, and who received the oral amoxicillin challenge
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Intent-to-Treat Population: All subjects who had valid skin testing performed (i.e., administered all components of the Penicillin Skin Test Kit and the histamine control results are valid) and who receive the oral amoxicillin challenge.
Arm/Group | Intent-to-Treat Population
Number analyzed (Participants) | 391
percentage of participants | 98.0 [96.6 to 99.4]

ADVERSE EVENTS:
Time Frame: Adverse events were recorded immediately following administration of the Penicillin Skin Test and throughout the 3-day study period as spontaneously reported by subjects, reported during the phone interview ≥72-hours post-oral challenge, or observed by the site staff.
Groups:
- Safety Population-All Study-Emergent Adverse Events; Subjects With AE Related to Oral Amox Challenge: Intervention: Penicillin skin test kit
  The skin test procedure first involved puncture testing. Subjects who had negative skin puncture test results to any of the drug antigens contained within the Penicillin Skin Test Kit then underwent intradermal testing in duplicate. Subjects who had any positive skin test to drug antigens in the Penicillin Skin Test Kit were asked to return in 4 weeks to confirm the positive test(s). Subjects who had negative puncture and intradermal test results were given the oral amoxicillin challenge, which was comprised of a single, age-dependent, full oral dose of amoxicillin. The purpose of the oral amoxicillin challenge was to confirm absence of allergy and confirm the NPV of skin testing. Subjects were monitored at the study site for 1 hour following oral amoxicillin challenge and then sent home. The study site followed up by telephone with all subjects ≥72 hours after administration of the oral amoxicillin challenge.
- Subjects With AE Related to Skin Testing: Intervention: Penicillin skin test kit
  The skin test procedure first involved puncture testing. Subjects who had negative skin puncture test results to any of the drug antigens contained within the Penicillin Skin Test Kit then underwent intradermal testing in duplicate. Subjects who had any positive skin test to drug antigens in the Penicillin Skin Test Kit were asked to return in 4 weeks to confirm the positive test(s).
Arm/Group | Safety Population-All Study-Emergent Adverse Events | Subjects With AE Related to Skin Testing | Subjects With AE Related to Oral Amox Challenge
Serious Adverse Events (participants affected / at risk) | 0/481 | 0/481 | 0/391
Other Adverse Events (participants affected / at risk) | 53/481 | 7/481 | 12/391
OTHER ADVERSE EVENTS (reported when occurring in more than 0.2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Safety Population-All Study-Emergent Adverse Events (N=481) | Subjects With AE Related to Skin Testing (N=481) | Subjects With AE Related to Oral Amox Challenge (N=391)
Pruritus (Skin and subcutaneous tissue disorders) | 15 | 2 | 2
Rash (Skin and subcutaneous tissue disorders) | 6 | 1 | 2
Post-procedural hematoma (Skin and subcutaneous tissue disorders) | 5 | 3 | 0
Erythema (Skin and subcutaneous tissue disorders) | 4 | 1 | 2
Diarrhea (Gastrointestinal disorders) | 4 | 0 | 2
Abdominal discomfort (Gastrointestinal disorders) | 3 | 0 | 2
Chest discomfort (General disorders) | 3 | 1 | 0
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 3 | 1 | 0
Flushing (Vascular disorders) | 3 | 1 | 2
Headache (Nervous system disorders) | 2 | 0 | 1
Pruritus generalised (Skin and subcutaneous tissue disorders) | 2 | 0 | 1
Rash pruritic (Skin and subcutaneous tissue disorders) | 2 | 0 | 1
Urticaria (Immune system disorders) | 2 | 1 | 1
Dermatitis (Skin and subcutaneous tissue disorders) | 1 | 0 | 1
Rash erythematous (Skin and subcutaneous tissue disorders) | 1 | 0 | 1
Rash macular (Skin and subcutaneous tissue disorders) | 1 | 0 | 1
Skin disorder (Skin and subcutaneous tissue disorders) | 1 | 0 | 1
Abdominal pain upper (Gastrointestinal disorders) | 1 | 0 | 1
Vomiting (Gastrointestinal disorders) | 1 | 0 | 1
Chills (General disorders) | 1 | 0 | 1
Oedema peripheral (General disorders) | 1 | 0 | 1
Pain (General disorders) | 1 | 0 | 1
Angiodema (Immune system disorders) | 1 | 0 | 1
Joint stiffness (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1
Respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No